CLINICAL TRIAL: NCT04832906
Title: Ulipristal Acetate Therapy Versus Uterine Artery Embolization in Management of Uterine Fibroids
Brief Title: UA Versus UAE in Treatment of Fibroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Paula Naseef, Principal Investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU M D 71/2019
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Uterine Fibroid
Keywords: Abnormal uterine bleeding (AUB); Benign gynecologic conditions; Ulipristal acetate; Uterine artery embolization
MeSH Terms: conditions — Leiomyoma; Metrorrhagia | interventions — ulipristal; Uterine Artery Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A "Ulipristal Acetate (UA) - Fibristal group" (n=35) (Active Comparator): Patients within this group received oral Ulipristal Acetate (Fibristal ©) 5 mg / day starting from the first day of menstrual bleeding, and for 3 months (period of the study).
  Interventions: Drug: Ulipristal Oral Tablet
- Group B "Uterine artery embolization (UAE) group" (n=35) (Active Comparator): Patients within this group underwent bilateral selective uterine artery embolization, during which polyvinyl alcohol (PVA) particles was administered via a catheter followed by capping with a plug of gelatin sponge. The end point for embolization is to have a static column of contrast in the uterine artery, with only a stump filling when the internal iliac artery was injected. The gelatin sponge cap was thought to both complete the occlusion of the uterine artery and to prevent PVA particles from being drawn out of the uterine artery by the Venturi effect, which would result in non-target embolization.
  Interventions: Procedure: Uterine artery embolization

INTERVENTIONS:
Drug: Ulipristal Oral Tablet — A selective progesterone receptor modulator (SPRM), as a medical line of treatment for uterine fibroids. Due to its selective anti-proliferative and pro-apoptotic action, Ulipristal Acetate (UA) is assumed to be effective in reducing abnormal uterine bleeding (AUB) and fibroid size.
  Arms: Group A "Ulipristal Acetate (UA) - Fibristal group" (n=35)
Procedure: Uterine artery embolization — Selective embolization of uterine arteries bilaterally, using polyvinyl alcohol (PVA) particles administered via a catheter followed by capping with a plug of gelatin sponge. The end point for embolization is to have a static column of contrast in the uterine artery, with only a stump filling when the internal iliac artery was injected.
  Arms: Group B "Uterine artery embolization (UAE) group" (n=35)

SUMMARY:
Study objective: To prove that Ulipristal acetate is an effective line of management for uterine fibroids by causing a significant decline in fibroid volumes resulting in a substantial relief of fibroid-related symptoms, and to compare its results with those of uterine artery embolization.

Design: A randomized control trial. Setting: Maternity Hospital, Ain Shams University.

Patients: Women with symptomatic uterine fibroids.

Interventions: 70 women were randomly assigned to either Ulipristal Acetate (UA) group or uterine artery embolization (UAE) group (35 in each group). Both groups were followed up to detect the decline in fibroid size as well as the improvement of symptoms.

DETAILED DESCRIPTION:
Inclusion Criteria:

Women with symptomatic uterine fibroids were recruited into the study after fulfilling the following criteria:

* Their age should range from 35 to 50 years.
* Their body mass index (BMI) should range from 18 to 35 Kg/m2.
* The presence of multiple symptomatic type 2, 3, 4, 5, or 6 uterine fibroids according to the FIGO classification.
* The dominant fibroid diameter should range from 4 to 8 cm as assessed by ultrasound.
* They should not be seeking future fertility.
* They should be refusing any surgical intervention whether myomectomy or hysterectomy.

Exclusion Criteria:

1. Post-menopausal status or premature ovarian failure.
2. Type 0, 1 and 7 uterine fibroids according to FIGO classification.
3. Previous myomectomy or any uterine surgery.
4. Previous or ongoing hormonal treatment.

Sampling Method:

The study sample will be a "convenient sample" where women fulfilling the inclusion criteria and consenting to participate in the study will be recruited.

Sample Size justification:

The study will include 70 women with symptomatic uterine fibroids who will be randomized into two groups with 35 women in each group.

The required sample size has been calculated using the PASS 15 Power Anal-ysis and Sample Size Software (PASS©) version 15 (2017); NCSS, LLC. Kaysville, Utah, USA.

The main outcome measure is the reduction in fibroid volume. The secondary outcome measures are symptoms relief and improvement in quality of life.

A previous study reported that Ulipristal Acetate (UA) was comparable to uterine artery embolization (UAE) as regards the percentage of reduction in fibroid volume with median (interquartile range) percentage reduction of 48.1 (24.8 - 66) % versus 47.3 (29.5 - 69.5) % for UPA and UAE respectively (Czuczwar et al., 2015).

Using the methods described by Wan et al (2014) and Luo et al (2018), we calculated that the mean ± SD percentage of reduction in fibroid volume was 44.0 ± 28.5 % versus 48.9 ±32.3 % for UPA and UAE respectively, with mean difference of 4.9 % and common within group SD of 30.5%.

Taking into consideration a "drop-out rate" of about 10%, due to loss of follow up or withdrawal from the study, it is estimated that a sample size of 35 patients per group achieves 80% power using a one-sided equivalence test with a significance level of 5% (alpha-error = 0.05), when the difference between the two means is 4.9 %, common within group SD is 30.5 %, and equivalence limits are -25% and 25%.

On the other hand, this sample size achieves a power of 82% to detect a statistically significant difference between the two groups as regards the symptoms scores and measures of ovarian reserve (AFC and AMH) for an effect size equivalent to a Cohen's d of 0.75 (i.e., 0.75 common SD) using a two-sided unpaired t-test with the same significance level of alpha = 0.05.

These equivalence limits and effect size have been targeted, as they may be considered clinically important.

Informed consent:

The nature and scope of the clinical study will be explained in an understand-able way to the patients and an informed consent form, in Arabic language, including all the study procedures, advantages and possible risks and specifying who informed the patient, will be provided and the patient must sign on it before participation. The study protocol and patient informed consent will be reviewed and approved by the Ethics Committee of the Obstetrics and Gynecology Department, Ain Shams University.

Funding:

This study will be funded by the researcher himself and Ain Shams University

Randomization and Allocation concealment:

The participants will be randomly assigned into one of the two study groups using a computer random sequence generator. The randomization will be made using sequentially numbered, opaque sealed envelopes; each envelope contains the method of intervention according to the random sequence and will be opened just before the intervention.

Study Procedures:

All participants will undergo full assessment before starting either treatment options. This assessment will include:

Detailed History:

* Personal history: including patient's full name, age, marital status, parity, occupation and residence will be recorded.
* Menstrual history: including age of menarche, D/C, amount of menstrual flow and associated dysmenorrhea.
* Contraceptive history: to exclude other causes for uterine bleeding.
* Past medical history of Diabetes Mellitus, hypertension, bronchial asthma, cardiac diseases, anemia, etc.
* Past surgical history of uterine surgeries.
* History of present illness with detailed analysis of each patient's complaint whether abnormal uterine bleeding, dysmenorrhea and pelvic pressure symptoms such as urinary urgency or constipation.

Physical Examination:

* General examination including: Pulse, blood pressure, temperature, body mass index (BMI), auscultation of lungs and heart, and complex-ion as pallor due to anemia caused by heavy bleeding.
* Abdominal examination: inspection for any scar, palpation of the abdomen for any tenderness and for pelviabdominal masses.
* Pelvic examination: complete bimanual examination for uterine size, mobility and palpable uterine fibroids.

Investigations:

* Baseline hemoglobin, hematocrit, and blood grouping.
* Blood chemistry: AST, ALT, serum creatinine and RBS.
* Trans-vaginal ultrasound for uterine volume and fibroid location, volume and maximum diameter. Uterine volume (expressed in cubic centimeters) will be calculated by measuring the maximum length, antero-posterior and transverse diameters of the uterine corpus, using the US device software formula for calculation of the uterine volume. Myoma volumes will be measured by using the existing 2-dimensional US methods. The FIGO classification system (figure 1) will be used for defining the myoma location.

Study groups:

Patients recruited in this study will be randomized into one of the following study groups:

1. Group A "Ulipristal Acetate (UA) - Fibristal group" (n=35):

   Patients within this group will receive oral Ulipristal Acetate (Fibristal ©) 5 mg / day starting from the first day of menstrual bleeding, and for 3 months (period of the study).
2. Group B "Uterine artery embolization (UAE) group" (n=35):

Patients within this group will undergo bilateral selective uterine artery embolization, during which polyvinyl alcohol (PVA) particles will be administered via a catheter followed by capping with a plug of gelatin sponge. The end point for embolization is to have a static column of contrast in the uterine artery, with only a stump filling when the internal iliac artery was injected. The gelatin sponge cap was thought to both complete the occlusion of the uterine artery and to prevent PVA particles from being drawn out of the uterine artery by the Venturi effect, which would result in non-target embolization.

Follow up:

Each patient within both groups will be subjected to follow-up trans-vaginal ultrasound (US) 3 months after Ulipristal acetate (UA) therapy or after uterine artery embolization (UAE) session to detect the decline in uterine fibroid volumes in comparison to their baseline. To reduce inter-observer variability associated with ultrasound imaging, measurements will be always taken by the same sonographer.

Each patient within both groups will be evaluated clinically for the symptoms reported at least 1 month before starting the treatment (baseline) and 3 months after Ulipristal acetate (UA) therapy or after uterine artery embolization (UAE) session. Durability of the used treatment line will be tested by follow up after one year from initiating therapy.

Fibroid-related heavy menstrual bleeding (HMB) will be evaluated by the pictorial blood assessment chart score (figure 2). This instrument is a self-administered pictorial chart that takes account of the number of sanitary pads and tampons used, presence of blood clots, and episodes of bleeding. The 1-month pictorial blood assessment chart score was calculated from the addition of daily scores for 28 days. A score of higher than 100 during the first 8 days of menstruation will be defined as heavy menstrual bleeding (HMB).

Subjective feelings of pelvic pressure, urinary urgency, and constipation will be recorded on a simplified questionnaire containing 2 categories defined as "absent "and "present." The visual analog scale (VAS) pain score (figure 3) will be used to determine the presence or absence of pelvic pain.

Statistical Methods:

Data will be analyzed using Intention to treat (ITT) analysis. According to Fisher et al (1990), the ITT analysis includes all randomized patients in the groups to which they were randomly assigned, regardless of their adherence with the entry criteria, regardless of the treatment they actually received, and regardless of subsequent withdrawal from treatment or deviation from the protocol.

In other words, ITT analysis includes every subject who is randomized according to randomized treatment assignment. It ignores non-compliance, protocol deviations, withdrawal, and anything that happens after randomization. ITT analysis is usually described as "once randomized, always analyzed".

ITT analysis avoids overoptimistic estimates of the efficacy of one of the two interventions resulting from the removal of non-compliers by accepting that noncompliance and protocol deviations are likely to occur in actual clinical practice.

Efficacy of the two study interventions will be compared using Odds ratio (OR), Relative risk (RR), Number needed to treat (NNT) and Number needed to harm (NNH).

Data will be analyzed using IBM© SPSS© Statistics version 23 (IBM© Corp., Armonk, NY). Normally distributed numerical data will be presented as mean and SD, and skewed data as median and interquartile range. Qualitative data will be presented as number and percentage. Normally distributed numerical data will be compared using the unpaired t test and skewed data using the Mann-Whitney test. Categorical data will be compared using the Pearson chi-squared test or Fisher's exact test, if appropriate. A two-sided p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Their age should range from 35 to 50 years.
* Their body mass index (BMI) should range from 18 to 35 Kg/m2.
* The presence of one or more symptomatic type 2, 3, 4, 5, or 6 uterine fibroids according to the FIGO classification.
* The dominant fibroid diameter should range from 4 to 8 cm as assessed by ultrasound.
* They should not be seeking future fertility.
* They should be refusing any surgical intervention whether myomectomy or hysterectomy.

Exclusion Criteria:

* Post-menopausal status or premature ovarian failure.
* Type 0, 1 and 7 uterine fibroids according to FIGO classification.
* Previous myomectomy or any uterine surgery.
* Previous or ongoing hormonal treatment.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Decline in dominant fibroid volume (in cubic centimeters). | 3 months
  measured by transvaginal ultrasound.

SECONDARY OUTCOMES:
Relief of abnormal uterine bleeding. | 3 months
  measured by reduction in Pictorial Blood Loss Assessment Chart Score.
Relief of pelvic pain. | 3 months
  measured by reduction in Visual Analogue Scale Score.
Relief of pelvic pressure symptoms. | 3 months
  Subjective feelings of pelvic pressure symptoms including urinary urgency, and constipation was recorded using a simplified questionnaire containing 2 categories defined as "absent "and "present."
Adverse effects. | 6 months
  resulting from either treatment options within the 2 arms of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No